CLINICAL TRIAL: NCT00421304
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate a Single Intravenous Dose of Motavizumab (MEDI-524), a Humanized Enhanced Potency Monoclonal Antibody Against Respiratory Syncytial Virus (RSV), for the Treatment of Children Hospitalized With RSV Illness
Brief Title: A Study to Evaluate a Single Intravenous Dose of Motavizumab for the Treatment of Children Hospitalized With Respiratory Syncytial Virus (RSV) Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP141
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Results first posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-07

CONDITIONS: RSV Illness in ≤12 Months of Participants
Keywords: Respiratory Syncytial Virus illness; RSV
MeSH Terms: interventions — motavizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive a single intravenous (IV) dose of placebo matched to motavizumab on Day 0 of the study.
  Interventions: Other: Placebo
- Motavizumab 30 mg/kg (Experimental): Participants will receive a single IV dose of motavizumab 30 mg/kg on Day 0 of the study.
  Interventions: Biological: Motavizumab
- Motavizumab 100 mg/kg (Experimental): Participants will receive a single IV dose of motavizumab 100 mg/kg on Day 0 of the study.
  Interventions: Biological: Motavizumab

INTERVENTIONS:
Biological: Motavizumab — A single IV dose of motavizumab 30 mg/kg or 100 mg/kg will be administered on Day 0 of the study.
  Other Names: MEDI-524
  Arms: Motavizumab 100 mg/kg; Motavizumab 30 mg/kg
Other: Placebo — A single IV dose of placebo matched to motavizumab will be administered on Day 0 of the study.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to describe the effect of a single dose of medication compared to placebo in the upper respiratory tract in previously healthy children less than or equal to 12 months of age who are hospitalized with lower respiratory tract illness.

DETAILED DESCRIPTION:
The primary objective of this study is to describe the effect of a single 30 mg/kg or 100 mg/kg intravenous (IV) dose of Motavizumab compared to placebo on study drug levels and viral load as measured by cultivatable virus and real-time reverse transcriptase-polymerase chain reaction (RT-PCR) in the upper respiratory tract in previously healthy children ≤12 months of age who are hospitalized with lower respiratory tract illness.

ELIGIBILITY:
Inclusion Criteria:

Children must meet all of the following criteria:

* Previously healthy
* Age less or equal to 12 months at the time of randomization
* Gestational age more or equal to 36 weeks
* Hospitalized for lower respiratory tract illness (i.e., RSV bronchiolitis and/or pneumonia)
* Documented positive RSV test within 48 hours prior to randomization
* Randomization within 12 hours of the decision to hospitalize a child for RSV illness
* Written informed consent obtained from the participant's parent(s)/legal guardian

Exclusion Criteria:

Children must have none of the following:

* Prior receipt of or receiving ribavirin or other anti-viral treatment for the current episode of RSV infection prior to randomization
* Any use of systemic or inhaled steroids within the past 30 days prior to randomization
* Intubation for ventilatory support at randomization
* Any medically significant underlying ongoing chronic illness or organ system dysfunction, or other known acute illness except for RSV infection
* Known renal impairment, hepatic dysfunction, hematologic abnormalities, seizure or other neurologic disorder or immunodeficiency
* Requirement for supplemental oxygen at any time prior to the current RSV infection (brief use of oxygen in the immediate postnatal period to treat a transient condition is allowed)
* Mechanical ventilation at any time prior to the onset of the current RSV infection
* Congenital heart disease [children with medically or surgically closed patent ductus arteriosis (PDA), small atrial septal defect (ASD) or small ventricular septal defect (VSD) will be allowed]
* Previous reaction to IVIG, blood products, or other foreign proteins
* Prior use of intravenous immunoglobulin (IVIG), palivizumab (SynagisÒ), or other immunoglobulin products within the past 2 months
* Currently receiving other investigational agents or have received any other investigational agents within the 3 months prior to randomization
* Prior or current participation in any investigational study with a therapeutic agent or vaccine for RSV

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2007-01-10 (Actual); Primary Completion 2009-09-17 (Actual); Study Completion 2009-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Pamela Griffin, M.D., Study Director — MedImmune LLC
Locations (33):
- United States (26):
  - Research Site, Tucson, Arizona
  - Research Site, Long Beach, California
  - Research Site, Orange, California
  - Research Site, San Diego, California
  - Research Site, Jacksonville, Florida
  - Research Site, Honolulu, Hawaii
  - Research Site, Chicago, Illinois
  - Research Site, Oak Lawn, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, Jackson, Mississippi
  - Research Site, Omaha, Nebraska
  - Research Site, Brooklyn, New York
  - Research Site, Buffalo, New York
  - Research Site, Mineola, New York
  - Research Site, New Hyde Park, New York
  - Research Site, Rochester, New York
  - Research Site, Syracuse, New York
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Seattle, Washington
  - Research Site, Morgantown, West Virginia
  - Research Site, Milwaukee, Wisconsin
- Research Site, Herston, Australia
- Chile (2):
  - Research Site, Independencia
  - Research Site, Santiago
- New Zealand (3):
  - Research Site, Auckland
  - Research Site, Hamilton
  - Research Site, Palmerston North
- Research Site, Panama City, Panama

REFERENCES:
- [Derived] Ramilo O, Lagos R, Saez-Llorens X, Suzich J, Wang CK, Jensen KM, Harris BS, Losonsky GA, Griffin MP; Motavizumab Study Group. Motavizumab treatment of infants hospitalized with respiratory syncytial virus infection does not decrease viral load or severity of illness. Pediatr Infect Dis J. 2014 Jul;33(7):703-9. doi: 10.1097/INF.0000000000000240. PMID 24356256

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received a single intravenous (IV) dose of placebo matched to motavizumab on Day 0 of the study.
- Motavizumab 30 mg/kg: Participants received a single IV dose of motavizumab 30 mg/kg on Day 0 of the study.
- Motavizumab 100 mg/kg: Participants received a single IV dose of motavizumab 100 mg/kg on Day 0 of the study.
Period: Overall Study
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Started | 40 | 39 | 39
Completed | 32 | 35 | 31
Not Completed | 8 | 4 | 8
Not completed — Lost to Follow-up | 5 | 2 | 5
Not completed — Withdrawal by Subject | 2 | 2 | 2
Not completed — Mistakenly randomized, chose not to participate in study | 1 | 0 | 0
Not completed — Did not attend Day 360 visit | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent to treat population (ITT) included all participants who were randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg | Total
Number analyzed (Participants) | 40 | 39 | 39 | 118
Age, Continuous [Mean (Standard Deviation); unit: Months] | 3.72 (2.90) | 3.07 (2.62) | 3.47 (2.98) | 3.42 (2.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 19 | 19 | 49
  Male | 29 | 20 | 20 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 35 | 32 | 96
  Not Hispanic or Latino | 11 | 4 | 7 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 5 | 2 | 2 | 9
  White | 26 | 26 | 27 | 79
  More than one race | 3 | 0 | 0 | 3
  Unknown or Not Reported | 5 | 10 | 9 | 24

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Syncytial Virus (RSV) Load in the Upper Respiratory Tract as Measured by Quantitative Real Time Reverse Transcriptase Polymerase Chain Reaction (RT-PCR) at Day 0
Description: The RSV viral load is measured by cultivatable virus and real-time RT-PCR in the upper respiratory tract in previously healthy children less than or equal to (<=12) months of age who are hospitalized with lower respiratory tract illness.
Time Frame: Day 0
Population: The ITT population included all participants who were randomized in the study. Participants with adequate baseline samples and who tested positive for RSV at Day 0 were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 37 | 39 | 36
log10 copies/mL | 8.13 (0.73) | 8.05 (1.22) | 8.15 (0.86)
Statistical Analysis 1: Comparison: Placebo vs Motavizumab 30 mg/kg; Test type: Superiority; p = 0.218, Wilcoxon's rank-sum test
Statistical Analysis 2: Comparison: Placebo vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.643, Wilcoxon's rank-sum test
Statistical Analysis 3: Comparison: Motavizumab 30 mg/kg vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.677, Wilcoxon's rank-sum test

2. Primary Outcome: RSV Load in the Upper Respiratory Tract as Measured by Quantitative RT-PCR at Day 1
Description: The RSV viral load is measured by cultivatable virus and real-time RT-PCR in the upper respiratory tract in previously healthy children <=12 months of age who are hospitalized with lower respiratory tract illness.
Time Frame: Day 1
Population: The ITT population included all participants who were randomized in the study. Participants with adequate baseline samples and who tested positive for RSV at Day 1 were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 37 | 38 | 36
log10 copies/mL | 7.61 (0.86) | 7.54 (1.26) | 7.40 (1.26)
Statistical Analysis 1: Comparison: Placebo vs Motavizumab 30 mg/kg; Test type: Superiority; p = 0.257, Wilcoxon's rank-sum test
Statistical Analysis 2: Comparison: Placebo vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.726, Wilcoxon's rank-sum test
Statistical Analysis 3: Comparison: Motavizumab 30 mg/kg vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.551, Wilcoxon's rank-sum test

3. Primary Outcome: RSV Load in the Upper Respiratory Tract as Measured by Quantitative RT-PCR at Day 2
Description: as for outcome 2
Time Frame: Day 2
Population: The ITT population included all participants who were randomized in the study. Participants with adequate baseline samples and who tested positive for RSV at Day 2 were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 37 | 38 | 36
log10 copies/mL | 6.95 (1.21) | 6.68 (1.21) | 6.59 (1.35)
Statistical Analysis 1: Comparison: Placebo vs Motavizumab 30 mg/kg; Test type: Superiority; p = 0.591, Wilcoxon's rank-sum test
Statistical Analysis 2: Comparison: Placebo vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.393, Wilcoxon's rank-sum test
Statistical Analysis 3: Comparison: Motavizumab 30 mg/kg vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.586, Wilcoxon's rank-sum test

4. Primary Outcome: RSV Load in the Upper Respiratory Tract as Measured by Quantitative RT-PCR at Day 3
Description: as for outcome 2
Time Frame: Day 3
Population: The ITT population included all participants who were randomized in the study. Participants with adequate baseline samples and who tested positive for RSV at Day 3 were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 34 | 38 | 32
log10 copies/mL | 6.12 (1.15) | 6.11 (1.26) | 5.95 (1.46)
Statistical Analysis 1: Comparison: Placebo vs Motavizumab 30 mg/kg; Test type: Superiority; p = 0.894, Wilcoxon's rank-sum test
Statistical Analysis 2: Comparison: Placebo vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.674, Wilcoxon's rank-sum test
Statistical Analysis 3: Comparison: Motavizumab 30 mg/kg vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.636, Wilcoxon's rank-sum test

5. Primary Outcome: RSV Load in the Upper Respiratory Tract as Measured by Quantitative RT-PCR at Day 4
Description: as for outcome 2
Time Frame: Day 4
Population: The ITT population included all participants who were randomized in the study. Participants with adequate baseline samples, who tested positive for RSV at Day 4 were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 10 | 10 | 15
log10 copies/mL | 6.00 (0.58) | 5.76 (0.82) | 5.41 (1.44)
Statistical Analysis 1: Comparison: Placebo vs Motavizumab 30 mg/kg; Test type: Superiority; p = 0.397, Wilcoxon's rank-sum test
Statistical Analysis 2: Comparison: Placebo vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.238, Wilcoxon's rank-sum test
Statistical Analysis 3: Comparison: Motavizumab 30 mg/kg vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.461, Wilcoxon's rank-sum test

6. Primary Outcome: RSV Load in the Upper Respiratory Tract as Measured by Quantitative RT-PCR at Day 5
Description: as for outcome 2
Time Frame: Day 5
Population: The ITT population included all participants who were randomized in the study. Participants with adequate baseline samples, who tested positive for RSV at Day 5 were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 9 | 8 | 8
log10 copies/mL | 5.52 (0.68) | 5.26 (1.20) | 5.31 (1.94)
Statistical Analysis 1: Comparison: Placebo vs Motavizumab 30 mg/kg; Test type: Superiority; p = 0.322, Wilcoxon's rank-sum test
Statistical Analysis 2: Comparison: Placebo vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.747, Wilcoxon's rank-sum test
Statistical Analysis 3: Comparison: Motavizumab 30 mg/kg vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.717, Wilcoxon's rank-sum test

7. Primary Outcome: RSV Load in the Upper Respiratory Tract as Measured by Quantitative RT-PCR at Day 6
Description: as for outcome 2
Time Frame: Day 6
Population: The ITT population included all participants who were randomized in the study. Participants with adequate baseline samples, who tested positive for RSV at Day 6 were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 5 | 5 | 5
log10 copies/mL | 5.63 (0.91) | 5.25 (1.58) | 5.60 (2.08)
Statistical Analysis 1: Comparison: Placebo vs Motavizumab 30 mg/kg; Test type: Superiority; p = 0.847, Wilcoxon's rank-sum test
Statistical Analysis 2: Comparison: Placebo vs Motavizumab 100 mg/kg; Test type: Superiority; p = 1.000, Wilcoxon's rank-sum test
Statistical Analysis 3: Comparison: Motavizumab 30 mg/kg vs Motavizumab 100 mg/kg; Test type: Superiority; p = 1.000, Wilcoxon's rank-sum test

8. Primary Outcome: RSV Load in the Upper Respiratory Tract as Measured by Quantitative RT-PCR at Day 7
Description: as for outcome 2
Time Frame: Day 7
Population: The ITT population included all participants who were randomized in the study. Participants with adequate baseline samples and who tested positive for RSV at Day 7 were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 35 | 37 | 36
log10 copies/mL | 4.86 (1.45) | 4.73 (1.27) | 4.52 (1.70)
Statistical Analysis 1: Comparison: Placebo vs Motavizumab 30 mg/kg; Test type: Superiority; p = 0.653, Wilcoxon's rank-sum test
Statistical Analysis 2: Comparison: Placebo vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.283, Wilcoxon's rank-sum test
Statistical Analysis 3: Comparison: Motavizumab 30 mg/kg vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.411, Wilcoxon's rank-sum test

9. Primary Outcome: RSV Load in the Upper Respiratory Tract as Measured by Quantitative RT-PCR at Day 30
Description: as for outcome 2
Time Frame: Day 30
Population: The ITT population included all participants who were randomized in the study. Participants with adequate baseline samples and who tested positive for RSV at Day 30 were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 35 | 37 | 34
log10 copies/mL | 3.03 (1.11) | 3.05 (1.33) | 2.96 (1.08)
Statistical Analysis 1: Comparison: Placebo vs Motavizumab 30 mg/kg; Test type: Superiority; p = 0.988, Wilcoxon's rank-sum test
Statistical Analysis 2: Comparison: Placebo vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.832, Wilcoxon's rank-sum test
Statistical Analysis 3: Comparison: Motavizumab 30 mg/kg vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.748, Wilcoxon's rank-sum test

10. Primary Outcome: RSV Load in the Upper Respiratory Tract as Measured by Quantitative RT-PCR at Day 90
Description: as for outcome 2
Time Frame: Day 90
Population: The ITT population included all participants who were randomized in the study. Participants with adequate baseline samples and who tested positive for RSV at Day 90 were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 33 | 37 | 34
log10 copies/mL | 2.66 (0.70) | 2.55 (0.29) | 2.50 (0.00)
Statistical Analysis 1: Comparison: Placebo vs Motavizumab 30 mg/kg; Test type: Superiority; p = 0.280, Wilcoxon's rank-sum test
Statistical Analysis 2: Comparison: Placebo vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.108, Wilcoxon's rank-sum test
Statistical Analysis 3: Comparison: Motavizumab 30 mg/kg vs Motavizumab 100 mg/kg; Test type: Superiority; p = 1.000, Wilcoxon's rank-sum test

11. Primary Outcome: RSV Load in the Upper Respiratory Tract as Measured by Quantitative RT-PCR at Day 180
Description: as for outcome 2
Time Frame: Day 180
Population: The ITT population included all participants who were randomized in the study. Participants with adequate baseline samples and who tested positive for RSV at Day 180 were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 32 | 35 | 32
log10 copies/mL | 2.68 (0.95) | 2.52 (0.09) | 2.50 (0.00)
Statistical Analysis 1: Comparison: Placebo vs Motavizumab 30 mg/kg; Test type: Superiority; p = 0.742, Wilcoxon's rank-sum test
Statistical Analysis 2: Comparison: Placebo vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.486, Wilcoxon's rank-sum test
Statistical Analysis 3: Comparison: Motavizumab 30 mg/kg vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.490, Wilcoxon's rank-sum test

12. Primary Outcome: Motavizumab Concentration in Nasal Wash Aspirates at Day 0
Description: Motavizumab concentration in nasal wash aspirates is reported.
Time Frame: Day 0
Population: Evaluable population for pharmacokinetics (PK) included all participants who received a full dose of study drug. Participants with adequate motavizumab concentration in nasal wash aspirates at Day 0 were analyzed for the outcome.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 38 | 38
ng/mL | 0.93 (5.72) | 0.00 (0.00)
Statistical Analysis 1: Comparison: Motavizumab 30 mg/kg vs Motavizumab 100 mg/kg; Test type: Superiority; p = 1.000, Wilcoxon's rank-sum test

13. Primary Outcome: Motavizumab Concentration in Nasal Wash Aspirates at Day 1
Description: Motavizumab concentration in nasal wash aspirates is reported.
Time Frame: Day 1
Population: Evaluable population for PK included all participants who received a full dose of study drug. Participants with adequate motavizumab concentration in nasal wash aspirates at Day 1 were analyzed for the outcome.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 38 | 38
ng/mL | 4673.3 (5397.4) | 10087 (10242)
Statistical Analysis 1: Comparison: Motavizumab 30 mg/kg vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.050, Wilcoxon's rank-sum test

14. Primary Outcome: Motavizumab Concentration in Nasal Wash Aspirates at Day 2
Description: Motavizumab concentration in nasal wash aspirates is reported.
Time Frame: Day 2
Population: Evaluable population for PK included all participants who received a full dose of study drug. Participants with adequate motavizumab concentration in nasal wash aspirates at Day 2 were analyzed for the outcome.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 38 | 38
ng/mL | 2341.2 (2928.4) | 7436.7 (10321)
Statistical Analysis 1: Comparison: Motavizumab 30 mg/kg vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.008, Wilcoxon's rank-sum test

15. Primary Outcome: Motavizumab Concentration in Nasal Wash Aspirates at Day 7
Description: Motavizumab concentration in nasal wash aspirates is reported.
Time Frame: Day 7
Population: Evaluable population for PK included all participants who received a full dose of study drug. Participants with adequate motavizumab concentration in nasal wash aspirates at Day 7 were analyzed for the outcome.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 37 | 38
ng/mL | 966.37 (1016.0) | 2464.2 (2788.0)
Statistical Analysis 1: Comparison: Motavizumab 30 mg/kg vs Motavizumab 100 mg/kg; Test type: Superiority; p = 0.012, Wilcoxon's rank-sum test

16. Primary Outcome: Motavizumab Concentration in Nasal Wash Aspirates at Day 30
Description: Motavizumab concentration in nasal wash aspirates is reported.
Time Frame: Day 30
Population: Evaluable population for PK included all participants who received a full dose of study drug. Participants with adequate motavizumab concentration in nasal wash aspirates at Day 30 were analyzed for the outcome.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 37 | 36
ng/mL | 431.21 (597.6) | 1934.5 (3055.6)
Statistical Analysis 1: Comparison: Motavizumab 30 mg/kg vs Motavizumab 100 mg/kg; Test type: Superiority; p < 0.001, Wilcoxon's rank-sum test

17. Secondary Outcome: Duration of RSV Hospitalization
Description: Duration of RSV hospitalization is reported.
Time Frame: From Randomization Day (Day 0) to Discharge Day (up to Day 30)
Population: RSV evaluable population included all participants who were RSV positive at Study Day 0 by real-time RT-PCR.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 37 | 39 | 36
Days | 3.55 (2.43) | 3.98 (3.01) | 4.46 (4.33)

18. Secondary Outcome: Respiratory Assessment Change Score (RACS) Derived From Baseline
Description: The RACS assesses changes in wheezing and retractions as measured by respiratory distress assessment instrument (RDAI) score and changes in respiratory rate. A RDAI score is a measure of the degree of severity of wheezing and retractions, with score range from 0 to 17; higher scores indicate more severe disease. Respiratory rate is summarized by raw scores and standardized change score. A change in respiratory rate of less than or equal to (<=) 5% from baseline is counted as a change of 0 units and a change in respiratory rate is assigned 1 point per each 10% change in the respiratory rate. The RACS is calculated as arithmetic sum of RDAI score change and of standardized respiratory rate change (for example, a child showing improvement who had a RDAI of -5 and a respiratory rate change of -2 would have a RACS score of -7). The RACS assessment does not have a minimum and/or maximum scale range. A decrease in RACS represents improvement, whereas an increase signifies deterioration.
Time Frame: Baseline (Day 0), Days 1, 2, 3, 7, and 30
Population: RSV evaluable population included all participants who were RSV positive at Study Day 0 by real-time RT-PCR. Here, 'Number Analyzed' denotes those participants who were evaluable at the specific time point.
Measure: Mean (Standard Deviation); unit: Units on a score
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 37 | 39 | 36
Units on a score
  Day 1: number analyzed (Participants) | 37 | 36 | 36
  Day 1 | -1.81 (5.05) | -1.36 (4.47) | -2.11 (4.58)
  Day 2: number analyzed (Participants) | 37 | 37 | 36
  Day 2 | -2.14 (5.20) | -3.51 (4.72) | -3.61 (5.02)
  Day 3: number analyzed (Participants) | 34 | 37 | 32
  Day 3 | -4.29 (5.45) | -5.49 (4.53) | -5.41 (5.11)
  Day 7: number analyzed (Participants) | 33 | 35 | 33
  Day 7 | -5.70 (5.40) | -6.94 (4.89) | -6.18 (5.23)
  Day 30: number analyzed (Participants) | 33 | 37 | 33
  Day 30 | -6.00 (5.51) | -7.14 (4.88) | -7.79 (4.01)

19. Secondary Outcome: Oxygen Saturation Level During RSV Hospitalization
Description: Oxygen saturation level during RSV hospitalization is reported.
Time Frame: Days 0, 1, 2, 3, 7, and 30
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Percentage of oxygen saturation
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 37 | 39 | 36
Percentage of oxygen saturation
  Day 0: number analyzed (Participants) | 37 | 38 | 36
  Day 0 | 96.8 (2.5) | 97.5 (1.9) | 97.1 (3.1)
  Day 1: number analyzed (Participants) | 37 | 37 | 36
  Day 1 | 97.3 (2.3) | 98.1 (1.6) | 97.2 (2.1)
  Day 2: number analyzed (Participants) | 36 | 38 | 36
  Day 2 | 96.9 (2.4) | 97.3 (2.1) | 97.5 (2.0)
  Day 3: number analyzed (Participants) | 32 | 37 | 32
  Day 3 | 97.7 (1.8) | 97.6 (1.7) | 97.4 (2.3)
  Day 7: number analyzed (Participants) | 30 | 33 | 33
  Day 7 | 97.6 (1.9) | 97.8 (1.4) | 97.6 (2.3)
  Day 30: number analyzed (Participants) | 31 | 36 | 33
  Day 30 | 97.9 (1.7) | 98.1 (1.8) | 98.5 (1.3)

20. Secondary Outcome: Heart Rate During RSV Hospitalization
Description: Heart rate during RSV hospitalization is reported.
Time Frame: Days 0, 1, 2, 3, 7, and 30
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 37 | 39 | 36
Beats per minute
  Day 0 | 148.6 (17.8) | 155.6 (19.5) | 157.6 (17.0)
  Day 1: number analyzed (Participants) | 37 | 37 | 36
  Day 1 | 146.0 (18.0) | 145.9 (14.6) | 145.9 (17.3)
  Day 2: number analyzed (Participants) | 37 | 38 | 36
  Day 2 | 141.2 (11.9) | 139.6 (15.1) | 136.6 (17.3)
  Day 3: number analyzed (Participants) | 34 | 38 | 31
  Day 3 | 138.6 (14.8) | 140.7 (14.8) | 143.3 (17.4)
  Day 7: number analyzed (Participants) | 33 | 36 | 33
  Day 7 | 139.6 (14.8) | 141.4 (20.2) | 143.5 (15.9)
  Day 30: number analyzed (Participants) | 33 | 37 | 32
  Day 30 | 139.6 (13.4) | 140.3 (13.8) | 137.1 (13.0)

21. Secondary Outcome: Respiratory Rate During RSV Hospitalization
Description: Respiratory rate during RSV hospitalization is reported.
Time Frame: Days 0, 1, 2, 3, 7, and 30
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 37 | 39 | 36
Breaths per minute
  Day 0 | 46.86 (10.20) | 49.28 (8.93) | 51.78 (11.28)
  Day 1: number analyzed (Participants) | 37 | 36 | 36
  Day 1 | 44.35 (11.88) | 48.67 (12.41) | 48.00 (14.13)
  Day 2: number analyzed (Participants) | 37 | 37 | 36
  Day 2 | 46.46 (9.05) | 41.89 (10.76) | 44.11 (11.77)
  Day 3: number analyzed (Participants) | 34 | 37 | 31
  Day 3 | 43.03 (9.28) | 40.54 (8.54) | 43.68 (10.81)
  Day 7: number analyzed (Participants) | 33 | 35 | 33
  Day 7 | 41.76 (9.06) | 40.14 (9.14) | 43.64 (11.06)
  Day 30: number analyzed (Participants) | 33 | 37 | 33
  Day 30 | 38.45 (6.73) | 41.11 (12.81) | 38.45 (6.53)

22. Secondary Outcome: Number of Participants With Supplemental Oxygen Use During RSV Hospitalization
Description: Number of participants with supplemental oxygen use during RSV hospitalization is reported.
Time Frame: From Randomization Day (Day 0) to Discharge Day (up to Day 30)
Population: RSV evaluable population included all participants who were RSV positive at Study Day 0 by real-time RT-PCR. Participants with hospitalization information available were analyzed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 37 | 38 | 36
Participants | 24 | 30 | 29

23. Secondary Outcome: Duration of Supplemental Oxygen Use During RSV Hospitalization
Description: Duration of supplemental oxygen use during RSV hospitalization is reported.
Time Frame: From Randomization Day (Day 0) to Discharge Day (up to Day 30)
Population: RSV evaluable population included all participants who were RSV positive at Study Day 0 by real-time RT-PCR. Participants who received supplemental oxygen during RSV hospitalization were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 24 | 30 | 29
Days | 3.5 (1.8) | 4.1 (2.8) | 4.4 (4.1)

24. Secondary Outcome: Number of Participants on Mechanical Ventilation During RSV Hospitalization
Description: Number of participants on mechanical ventilation during RSV hospitalization is reported.
Time Frame: From Randomization Day (Day 0) to Discharge Day (up to Day 30)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 37 | 38 | 36
Participants | 0 | 2 | 2

25. Secondary Outcome: Duration of Mechanical Ventilation During RSV Hospitalization
Description: Duration of mechanical ventilation during RSV hospitalization is reported.
Time Frame: From Randomization Day (Day 0) to Discharge Day (up to Day 30)
Population: RSV evaluable population included all participants who were RSV positive at Study Day 0 by real-time RT-PCR. Participants who received mechanical ventilation during RSV hospitalization were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 0 | 2 | 2
Days |  | 7.81 (0.88) | 4.64 (2.30)

26. Secondary Outcome: Number of Participants Admitted to the Intensive Care Unit (ICU)
Description: Number of participants admitted to ICU is reported.
Time Frame: From Randomization Day (Day 0) to Discharge Day (up to Day 30)
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 37 | 38 | 36
Participants | 0 | 3 | 3

27. Secondary Outcome: Duration of ICU Stay During RSV Hospitalization
Description: Duration of ICU stay during RSV hospitalization is reported.
Time Frame: From Randomization Day (Day 0) to Discharge Day (up to Day 30)
Population: RSV evaluable population included all participants who were RSV positive at Study Day 0 by real-time RT-PCR. Participants who were admitted to ICU were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 0 | 3 | 3
Days |  | 7.3 (4.6) | 5.0 (4.0)

28. Secondary Outcome: Number of Participants With Medically-attended Wheezing Episodes
Description: Wheezing episodes are considered medically-attended wheezing episodes if the medical care provider verifies and documents wheezing in the medical record or, in the case of hospitalization, the medical care provider assigns a discharge diagnosis of asthma, bronchiolitis, wheezing, or reactive airway disease. A new wheezing episode is the one that occurs for more than 2 weeks after the diagnosis of the previous episode and the medical opinion is that the wheezing does not represent a persistence of the previous episode. Medically-attended wheezing episodes were calculated and reported in the range of 0 to 9 events.
Time Frame: From randomization (Day 0) through Day 360 (approximately 12 months)
Population: RSV evaluable population included all participants who were RSV positive at Study Day 0 by real-time RT-PCR.
Measure: Number; unit: Participants
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 37 | 39 | 36
Participants
  0 event | 2 | 0 | 2
  1 event | 19 | 20 | 18
  2 events | 9 | 6 | 7
  3 events | 1 | 4 | 4
  4 events | 2 | 4 | 3
  5 events | 2 | 3 | 2
  6 events | 2 | 1 | 0
  7 events | 0 | 0 | 0
  8 events | 0 | 0 | 0
  9 events | 0 | 1 | 0

29. Secondary Outcome: Serum Concentration of Motavizumab
Description: Motavizumab concentration in serum is reported.
Time Frame: Days 1, 7, 90, 180, and 360
Population: Evaluable population for PK included all participants who received a full dose of study drug. Participants with adequate motavizumab concentration in serum at the specified time points were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 38 | 38
mcg/mL
  Day 1: number analyzed (Participants) | 37 | 37
  Day 1 | 298.73 (88.99) | 863.05 (240.28)
  Day 7: number analyzed (Participants) | 24 | 25
  Day 7 | 192.87 (57.07) | 640.36 (95.69)
  Day 90: number analyzed (Participants) | 37 | 35
  Day 90 | 11.39 (9.35) | 30.81 (23.63)
  Day 180: number analyzed (Participants) | 34 | 31
  Day 180 | 0.64 (1.41) | 2.45 (3.54)
  Day 360: number analyzed (Participants) | 35 | 30
  Day 360 | 0.04 (0.26) | 0 (0)

30. Secondary Outcome: Number of Participants With Detectable Anti-motavizumab Antibodies
Description: Number of participants with detectable anti-motavizumab antibodies are reported. Detection is defined as an anti-motavizumab antibody titer with a dilution value of 1:30 or greater.
Time Frame: Days 0, 180, and 360
Population: Evaluable population for anti-drug antibody included all participants who received a full dose of study drug. Participants with adequate anti-motavizumab antibody titer samples at the specified time points were analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 38 | 38
Participants
  Day 0: number analyzed (Participants) | 36 | 38
  Day 0 | 1 | 1
  Day 180: number analyzed (Participants) | 34 | 31
  Day 180 | 11 | 10
  Day 360: number analyzed (Participants) | 35 | 30
  Day 360 | 21 | 14

31. Secondary Outcome: Change From Baseline in Serum Cytokine Levels
Time Frame: Baseline (Day 0, pre-dose) through Day 360
Population: RSV evaluable population included all participants who were RSV positive at Study Day 0 by real-time RT-PCR. Participants with adequate cytokine levels were analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: Picograms per millilitre (pg/mL)
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 30 | 34 | 28
Picograms per millilitre (pg/mL)
  Interleukin-1(IL-1) beta: Day 360 | -3.005 (12.043) | 0.48 (2.442) | 48.943 (236.734)
  IL-1 receptor antagonist (RA): Day 360 | -266.925 (502.650) | -107.834 (201.740) | -171.278 (599.988)
  IL-2: Day 360 | -7.881 (30.340) | 0.446 (7.604) | 108.245 (445.422)
  IL4: Day 360 | -0.717 (5.733) | 2.187 (8.596) | 5.394 (30.426)
  Il-5: Day 360 | 1.045 (4.661) | 0.763 (1.817) | 0.774 (8.296)
  IL-6: Day 360 | -41.180 (72.120) | -24.305 (61.462) | 118.469 (524.680)
  IL-7: Day 360 | -1.328 (7.797) | 0.691 (5.094) | 4.305 (36.131)
  IL-8: Day 360 | -20.059 (19.790) | -18.323 (25.204) | -21.440 (20.033)
  IL-9: Day 360 | 58.378 (308.184) | -45.673 (188.920) | -48.034 (204.545)
  IL-10: Day 360 | -11.407 (21.458) | -6.924 (7.927) | 3.786 (75.604)
  IL12 P70: Day 360 | -10.633 (49.320) | 2.660 (18.759) | 48.765 (239.216)
  IL13: Day 360 | -0.779 (8.086) | 1.744 (3.244) | 9.893 (54.188)
  IL-15: Day 360 | -4.999 (14.377) | -0.402 (1.473) | 33.618 (139.355)
  IL-17: Day 360 | 2.067 (16.207) | 8.056 (24.954) | 1.092 (22.159)
  Eotaxin: Day 360 | -8.790 (138.692) | 36.955 (118.098) | 202.122 (728.741)
  Basic fibroblast growth factor: Day (D) 360 | 1.886 (34.663) | -1.342 (6.920) | 6.593 (34.509)
  Granulocyte-colony stimulating factor (G-CSF):D360 | -98.351 (192.339) | -91.782 (184.339) | -42.870 (108.678)
  Granulocyte macrophage -CSF: Day 360 | -54.862 (185.534) | -7.439 (26.842) | 964.242 (4386.145)
  Interferon (IFN) gamma: Day 360 | -65.424 (258.871) | 9.164 (91.580) | 464.277 (2027.072)
  IFN alpha: Day 360 | -23.980 (121.625) | 12.281 (67.767) | 194.351 (835.999)
  IFN gamma induced protein 10 (IP-10): Day 360 | -1089.184 (1711.708) | -1028.280 (1105.987) | -460.829 (2216.789)
  Monocyte chemoattractant protein-1: Day 360 | -75.818 (96.097) | -52.910 (84.827) | 17.128 (376.408)
  Macrophage inflammatory protein (MIP)-1 alpha:D360 | 0.604 (7.309) | 0.689 (2.485) | -31.042 (182.639)
  MIP-1 beta: Day 360 | -1.950 (105.553) | 43.061 (121.617) | -1.354 (235.052)
  Platelet-derived growth factor (PDGF)-BB: Day 360 | 3461.665 (5874.913) | 4377.256 (6050.996) | 3631.464 (9603.609)
  Rantes: Day 360 | 783.389 (2664.670) | 2946.934 (8074.666) | 793.431 (2672.889)
  Tumor necrosis factor (TNF) alpha: Day 360 | -17.112 (62.119) | -2.676 (29.385) | 403.443 (1918.152)
  Vascular endothelial growth factor (VEGF): Day 360 | -17.908 (135.254) | -33.293 (125.224) | -39.069 (87.616)
  Monokine induced by gamma(MIG): Day 360 | 1046.002 (2735.420) | 1086.786 (1246.951) | 2465.946 (7714.076)

32. Secondary Outcome: Change From Baseline in Upper Respiratory Tract (Nasal Wash) Cytokine Levels
Description: Change from baseline in upper respiratory tract (nasal wash) cytokine levels are reported.
Time Frame: Baseline (Day 0, pre-dose) through Day 180
Population: RSV evaluable population included all participants who were RSV positive at Study Day 0 by real-time RT-PCR. Participants with adequate nasal wash cytokine levels at specified time points were analysed for this outcome.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 32 | 35 | 32
pg/mL
  IL-1 beta: Day 180 | -2607.852 (6378.263) | -2575.906 (3423.519) | -1772.376 (3150.626)
  IL-1 RA: Day 180 | -91761.764 (268797.553) | -97050.821 (200487.750) | -69391.250 (127840.986)
  IL-2: Day 180 | -0.849 (14.116) | -1.215 (10.959) | -0.458 (9.316)
  IL-4: Day 180 | -1.761 (3.090) | -1.897 (2.939) | -1.435 (3.571)
  IL-5: Day 180 | -0.077 (1.865) | -0.351 (7.077) | 1.732 (7.974)
  IL-6: Day 180 | -1139.081 (1061.467) | -930.388 (1730.515) | -551.482 (676.661)
  IL-7: Day 180 | -6.553 (26.065) | -20.954 (48.390) | -18.219 (58.020)
  IL-8: Day 180 | -26762.935 (83539.520) | -20794.797 (30409.576) | -8610.260 (14715.271)
  IL-9: Day 180 | -32.899 (40.569) | -48.923 (57.492) | -45.623 (85.438)
  Il-10: Day 180 | -55.412 (65.437) | -65.522 (107.589) | -37.755 (60.765)
  IL-12 P70: Day 180 | -52.927 (60.597) | -54.300 (55.463) | -40.912 (64.739)
  IL-13: Day 180 | -54.573 (151.800) | -59.583 (116.696) | -43.758 (93.016)
  IL-15: Day 180 | -4.018 (17.009) | -7.107 (14.202) | -5.039 (15.169)
  IL-17: Day 180 | -22.557 (27.252) | -31.352 (25.301) | -25.215 (36.297)
  Eotaxin: Day180 | -16.905 (140.534) | -42.034 (90.948) | -23.358 (78.999)
  Basic FGF: Day 180 | -82.364 (125.246) | -149.153 (267.861) | -117.656 (183.542)
  G-CSF:Day 180 | -3547.084 (7428.810) | -3732.054 (9873.369) | -112.012 (9701.760)
  GM-CSF: Day 180 | -86.359 (139.214) | -79.592 (119.261) | -79.668 (157.497)
  IFN gamma: Day180 | -5754.670 (27853.042) | -3026.337 (13551.380) | -2755.333 (15534.906)
  IFN alpha: Day180: number analyzed (Participants) | 32 | 35 | 31
  IFN alpha: Day180 | -59.346 (413.227) | -95.529 (442.959) | -15.090 (240.549)
  IP-10: Day 180 | 2907.151 (14396.032) | -21562.675 (94358.228) | -15729.066 (93210.658)
  MCP-1: Day 180 | -510.596 (821.385) | -336.373 (230.303) | -317.251 (532.157)
  MIP-1 alpha: Day 180 | -81.063 (106.178) | -79.610 (100.858) | -54.416 (96.391)
  MIP-1 beta: Day 180 | -924.715 (913.488) | -921.287 (770.658) | -824.330 (1063.855)
  PDGF-BB: Day 180 | -95.616 (197.836) | -90.821 (192.864) | -55.547 (127.111)
  Rantes: Day 180 | -244.749 (971.092) | -789.419 (3136.828) | -194.783 (493.671)
  TNF alpha: Day 180 | -1489.621 (3190.856) | -1038.889 (1660.820) | -610.185 (1129.565)
  VEGF: Day 180 | -1167.204 (1698.618) | -1118.459 (1365.524) | -700.258 (1154.582)
  MIG: Day 180 | -42371.446 (124818.988) | -6693.146 (25633.807) | -25881.359 (110834.744)

33. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: From the start of study drug (Day 0) through Day 90
Population: Safety population included all the participants who received any dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 37 | 38 | 38
Participants
  Any TEAEs | 33 | 28 | 32
  Any TESAEs | 6 | 6 | 7

34. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities Reported as TEAEs
Time Frame: From the start of study drug (Day 0) through Day 30
Population: Safety population included all the participants who received any dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
Number analyzed (Participants) | 37 | 38 | 38
Participants
  Hypoalbuminaemia | 0 | 1 | 0
  Blood urea increased | 0 | 0 | 1
  Liver function test abnormal | 0 | 1 | 0
  Anaemia | 1 | 3 | 1
  Thrombocythaemia | 1 | 0 | 1
  Platelet count increased | 0 | 1 | 0
  Hypokalaemia | 0 | 1 | 1
  Hypercalcaemia | 0 | 1 | 0
  Hyperkalaemia | 0 | 1 | 0
  Hypernatraemia | 1 | 0 | 0
  Hyperphosphatasaemia | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the start of study drug (Day 0) through Day 90
Description: Adverse events were reported for safety population. Safety population included all the participants who received any dose of study drug.
Arm/Group | Placebo | Motavizumab 30 mg/kg | Motavizumab 100 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 6/37 | 6/38 | 7/38
Other Adverse Events (participants affected / at risk) | 30/37 | 22/38 | 24/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=37) | Motavizumab 30 mg/kg (N=38) | Motavizumab 100 mg/kg (N=38)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=37) | Motavizumab 30 mg/kg (N=38) | Motavizumab 100 mg/kg (N=38)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 3 (3) | 1 (1)
Conjunctivitis (Eye disorders) | 3 (3) | 2 (2) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 4 (4) | 3 (3)
Vomiting (Gastrointestinal disorders) | 5 (6) | 4 (4) | 2 (2)
Bronchitis (Infections and infestations) | 9 (14) | 4 (6) | 5 (7)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 10 (10) | 6 (7) | 6 (7)
Nasopharyngitis (Infections and infestations) | 2 (2) | 8 (10) | 4 (4)
Otitis media (Infections and infestations) | 4 (4) | 2 (2) | 4 (4)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 3 (4)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction in not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.